CLINICAL TRIAL: NCT06504524
Title: Comparative Effectiveness of Elranatamab (PF 06863135) in Clinical Study C1071003 Versus Standard of Care (SOC) in a Real-World (RW) External Control Arm of Patients With Triple-Class Refractory (TCR) Multiple Myeloma (MM) From TherapyMonitor MM Germany
Brief Title: A Study to Compare the Effects of Elranatamab (PF 06863135) Versus Standard of Care (SOC) in Patients With Multiple Myeloma (MM) in Germany and US
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: C1071035; NCT06504524 (Registry Identifier: ClinicalTrials.gov)
Record Dates: First submitted 2024-06-24; First posted 2024-07-16 (Actual); Results first posted 2025-06-27 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-05

CONDITIONS: Multiple Myeloma
Keywords: Myeloma; Multiple Myeloma; relapsed Multiple Myeloma; refractory Multiple Myeloma; PF-06863135; BCMA; bispecific; bispecific antibody; BCMA-CD3 bispecific; Elranatamab; MagnetisMM-3; External Control Arm
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell | interventions — Standard of Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Elranatamab: Patient cohort treated with elranatamab, coming form clinical trial Magnetis MM-3 trial
  Interventions: Drug: Elranatamab
- Standard-of-care: Patients treated with the standard-of-care therapies according to G-BA's definition will come from real-world data sources
  Interventions: Drug: Standard of Care

INTERVENTIONS:
Drug: Elranatamab — BCMA-CD3 bispecific antibody
  Other Names: Elrexfio (brand name)
  Groups: Elranatamab
Drug: Standard of Care — control arm
  Groups: Standard-of-care

SUMMARY:
The purpose of the study is to understand how well elranatamab (PF-06863135) may be used for relapsed refractory multiple myeloma (RRMM). MM is a type of cancer that begins in plasma cells (white blood cells that produce antibodies). Sometimes MM might improve at first, but then gets resistant to the treatment and starts growing again (known as relapsed refractory).

This study medicine will be compared with standard-of-care (SOC) therapies. SOC are treatments that are accepted by medical experts as a proper treatment for a certain type of disease and that are widely used by doctors in real world.

For people receiving elranatamab, the study doctors will use data from the other clinical trial (MagnetisMM-3). The study doctors will also use data from multiplemany real-world sources (TherapyMonitor MM Germany and Flatiron Health), for SOC in clinical practice. This study does not seek any participants for enrollment.

The study doctors will compare the experiences of people receiving elranatamab to people receiving SOC therapies. This way, it will help the study doctors to know how well elranatamab can be used for RRMM treatment.

DETAILED DESCRIPTION:
This study aims to contextualize the outcomes of Study C1071003 by comparing a priori specified clinical effectiveness of patients treated with elranatamab using patient-level data from study C1071003 vs. RW external control of patients with TCE MM treated with SOC therapies from the TM-MM Germany dataset and from the Flatiron Health database. The study is an extension of studies C1071024 and C1071031 with more recent data and an alternative set of therapies included in the ECA, following the G-BA's definition of the appropriate comparator therapy, and with an alternative data base focusing on German patients. Effectiveness will be measured by Overall Survival, Progression-free Survival with no differentiation between primary and secondary endpoints. To further reduce the potential for bias, appropriate comparative effectiveness methods and statistical techniques will be utilized (propensity score weighting/matching methods and multivariable regression). If appropriate, multiple imputation by chained equations will be performed. No formal sample size estimations have been performed for this observational study.

All patients who meet the inclusion/exclusion criteria of the external control arm will be included in the analyses

This is a retrospective study, so issues of quality control at study sites, e.g., data queries, do not apply. Analyses are programmed according to the specifications in the protocol. . Statistical programming code and summary output will be reviewed by the study team, including a biostatistician, for accuracy and completeness. Final deliverables will be reviewed and verified by a second, independent analyst. All quality checks will be documented.

For the secondary data collected by the TM-MM Germany project, the completeness and plausibility checks have been carried out in three stages during the generation of the dataset include:

1. Online check during data entry (incomplete and non-plausible data entries trigger an error message)
2. Central individual review after completion of data entry by the TNXO team of clinical monitors (in-complete or non-plausible data entry triggers a query process).
3. Central review of data sets by the TNXO team of data analysts to find and exclude any duplicated patients

After the duplicate records are excluded, only complete and plausible records are included in the database. Once the TM-MM dataset is provided by TNXO to Cytel and Pfizer approves data access for Study C1071003, the study data management will adhere to pre-defined process guidelines, which mainly consist of data validation based on computer-assisted checking of variables/values. In the RW dataset, patients with any implausible/counter-intuitive data will be excluded from the sample during the selection of the study population or for the analysis of specific outcomes, as applicable. The study team will maintain adequate and accurate records to enable the conduct of the study to be fully documented.

The Flatiron databases are compliant with both the spirit and the letter of the Health Insurance Portability and Accountability Act of 1996 (HIPAA). The databases meet the criteria for a limited-use dataset and contain none of the data elements prohibited by HIPAA for limited-use datasets.

ELIGIBILITY:
Inclusion Criteria:

Aged 18 years and older at index date

Diagnosis of MM

Measurable disease according to IMWG criteria

ECOG performance status ≤2

Refractory to at least 1 proteasome inhibitor, 1 immunomodulatory drug, and 1 anti-CD38 treatment (ie, triple-class refractory [TCR])

At least 1 treatment according to G-BA's definition of standard of care following their TCR eligibility

Exclusion Criteria:

Acute plasma cell leukemia

Amyloidosis

Smoldering MM

Stem cell transplant within 12 weeks of index or active graft versus host disease (GVHD)

Active malignancy within 3 years before index, except for basal cell or squamous cell skin cancer or carcinoma in situ

Administration with an investigational drug within 30 days prior to index

1st treatment following TCR eligibility not according to G-BA's definition of standard of care

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated with elranatamab will come from the MagnetisMM-3 trial. Patients treated with the standard-of-care therapies according to G-BA's definition will come from real-world data sources.
Sampling Method: Non-Probability Sample
Enrollment: 633 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (2):
- Pfizer, New York, New York, United States
- Pfizer, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C1071035

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Data of eligible participants with triple class refractory (TCR) multiple myeloma (MM) treated with elranatamab [data utilized form clinical trial C1071003] or standard of care treatment (SOC) [data utilized from real world data (RWD) sources Therapy Monitor MM (TM-MM) Germany dataset and the Flatiron Health database] was collected.
Pre-assignment Details: Available data from eligible participants was evaluated in approximately 9 months (study start date: 01-September-2023 to study completion date: 31-May-2024) of this retrospective, observational study as per its objectives.
Groups:
- C1071003 Cohort A: Eligible participants with TCR-MM, who were B-cell maturation antigen (BCMA) naïve, who initiated elranatamab (PF-06863135) following TCR eligibility in study C1071003 (NCT04649359) Cohort A were included.
- RWD: TM-MM Database: Eligible participants with TCR-MM who initiated SOC treatment and were identified from TM-MM database in real world setting under routine clinical practice outside of clinical trials were included. This arm served as external control arm.
- RWD: Flatiron Health Database: Eligible participants with TCR-MM who initiated SOC treatment and were identified from Flatiron Health database in real world setting under routine clinical practice outside of clinical trials were included. This arm served as external control arm.
Period: Overall Study
Arm/Group | C1071003 Cohort A | RWD: TM-MM Database | RWD: Flatiron Health Database
Started | 118 | 277 | 238
Completed | 118 | 277 | 238
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- C1071003 Cohort A: Eligible participants with TCR-MM, who were BCMA naïve, who initiated elranatamab (PF-06863135) following TCR eligibility in study C1071003 (NCT04649359) Cohort A were included.
- Total: Total of all reporting groups
Arm/Group | C1071003 Cohort A | RWD: TM-MM Database | RWD: Flatiron Health Database | Total
Number analyzed (Participants) | 118 | 277 | 238 | 633
Age, Customized [Count of Participants; unit: Participants]
  Age: <65 years | 41 | 33 | 71 | 145
  Age: 65-74 years | 55 | 134 | 90 | 279
  Age: >=75 years | 22 | 110 | 77 | 209
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53 | 107 | 118 | 278
  Male | 65 | 170 | 120 | 355
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS): C1071003 Cohort A Versus TM-MM Database Using Inverse Probability of Treatment Weights (IPTW) Analysis
Description: OS: A) C1071003 Cohort A: OS was defined as time from the date of the first dose of elranatamab until death due to any cause. Participants were censored at loss to or end of follow-up. B) TM-MM Database: OS was defined as time from initiation of SOC until death due to any cause. Participants were censored at loss to follow-up or end of the study period. Kaplan Meier method was used for analysis. Retrospective data was evaluated in this observational study for approximately 9 months.
Time Frame: C1071003: First dose to death due to any cause or censoring whichever occurred first (maximum [max] follow-up of 2.09 years [Y]); TM-MM Database: SOC to death due to any cause or censoring whichever occurred first (max follow-up of 4.22Y)
Population: Eligible participants whose data was retrieved and was used in this retrospective cohort study. In this outcome measure, IPTW analysis was applied. IPTW eliminated the effect of confounding by observed baseline participant characteristics, improve covariate balance, and thereby obtained unbiased estimates of treatment effects.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | C1071003 Cohort A | RWD: TM-MM Database
Number analyzed (Participants) | 118 | 277
Months | 13.27 [9.59 to NA] — Upper limit of 95% confidence interval (CI) could not be estimated due to insufficient number of participants with events. | 14.29 [12.98 to 24.08]
Statistical Analysis 1: Comparison: C1071003 Cohort A vs RWD: TM-MM Database; Test type: Other; p = 0.615, Regression, Cox; Hazard Ratio (HR) = 1.128, 95% CI 2-sided [0.705 to 1.804] — IPTW hazard ratio (HR) were estimated using weighted Cox proportional hazard models and confidence intervals were estimated using robust error variances. Stabilized IPT weights truncated at the 99.5th percentile were used

2. Primary Outcome: OS: C1071003 Cohort A Versus Flatiron Health Database Using IPTW Analysis
Description: OS: A) C1071003 Cohort A: OS was defined as time from the date of the first dose of elranatamab until death due to any cause. Participants were censored at loss to or end of follow-up. B) Flatiron Health Database: OS was defined as time from initiation of SOC until death due to any cause. Participants were censored at loss to follow-up or end of the study period. Kaplan Meier method was used for analysis. Retrospective data was evaluated in this observational study for approximately 9 months.
Time Frame: C1071003: First dose to death due to any cause or censoring whichever occurred first (max follow-up of 2.09Y); Flatiron Health Database: SOC to death due to any cause or censoring whichever occurred first (max follow-up of 6.45Y)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | C1071003 Cohort A | RWD: Flatiron Health Database
Number analyzed (Participants) | 118 | 238
Months | 14.62 [9.59 to NA] — Upper limit of 95% CI could not be estimated due to insufficient number of participants with events. | 18.99 [13.14 to 24.74]
Statistical Analysis 1: Comparison: C1071003 Cohort A vs RWD: Flatiron Health Database; Test type: Other; p = 0.4429, Regression, Cox; Hazard Ratio (HR) = 1.18, 95% CI 2-sided [0.85 to 1.64] — IPTW HR were estimated using weighted Cox proportional hazard models and confidence intervals were estimated using robust error variances. Stabilized IPT weights truncated at the 99.5th percentile were used

3. Secondary Outcome: Progression Free Survival (PFS): C1071003 Cohort A Versus TM-MM Database Using IPTW Analysis
Description: PFS: A) C1071003 Cohort A: time from date of first dose of elranatamab until confirmed progressive disease (PD) per IMWG criteria or death due to any cause, whichever occurred first. Participants censored at loss to or end of follow-up. B) TM-MM Database: time from SOC to either date of progression or death due to any cause. Participants censored at loss to follow-up or end of study period. PD per IMWG criteria: increase of >=25% from lowest response value in any 1 or more of the criteria: serum protein electrophoresis test (SPEP) with absolute increase >0.5 g/dL; 24-hour urine protein electrophoresis (UPEP) with absolute increase >200 mg/24 h; in participants without measurable serum & urine M-protein, absolute increase of >10 mg/dL in difference between involved & uninvolved free light chains (FLC) level; or absolute bone marrow plasma cell percentage >10%. Kaplan Meier method used for analysis. Retrospective data evaluated in this observational study for approximately 9 months.
Time Frame: C1071003: First dose to PD or death due to any cause or censoring whichever occurred first (max follow-up of 2.09Y); TM-MM Database: SOC to PD or death due to any cause or censoring whichever occurred first (max follow-up of 4.22Y)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | C1071003 Cohort A | RWD: TM-MM Database
Number analyzed (Participants) | 118 | 277
Months | 13.01 [7.66 to NA] — Upper limit of 95% CI could not be estimated due to insufficient number of participants with events. | 9.00 [7.20 to 11.63]
Statistical Analysis 1: Comparison: C1071003 Cohort A vs RWD: TM-MM Database; Test type: Other; p = 0.120, Regression, Cox; Hazard Ratio (HR) = 0.66, 95% CI 2-sided [0.390 to 1.115] — [estimate comment as in outcome 2, analysis 1]

4. Secondary Outcome: PFS: C1071003 Cohort A Versus Flatiron Health Database Using IPTW Analysis
Description: PFS: A) C1071003 Cohort A: time from date of first dose of elranatamab until confirmed PD per IMWG criteria or death due to any cause, whichever occurred first. Participants censored at loss to or end of follow-up. B) Flatiron Health Database: time from SOC to either date of progression or death due to any cause. Participants censored at loss to follow-up or end of study period. PD per IMWG criteria: increase of >=25% from lowest response value in any 1 or more of the criteria: SPEP with absolute increase >0.5 g/dL; 24-hour UPEP with absolute increase >200 mg/24 h; in participants without measurable serum and urine M-protein, absolute increase of >10 mg/dL in difference between involved and uninvolved FLC level; or absolute bone marrow plasma cell percentage >10%. Kaplan Meier method used for analysis. Retrospective data evaluated in this observational study for approximately 9 months.
Time Frame: C1071003: First dose to PD or death due to any cause or censoring whichever occurred first (max follow-up of 2.09Y); Flatiron Health Database: SOC to PD or death due to any cause or censoring whichever occurred first (max follow-up of 6.45Y)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | C1071003 Cohort A | RWD: Flatiron Health Database
Number analyzed (Participants) | 118 | 238
Months | 10.58 [3.42 to NA] — Upper limit of 95% CI could not be estimated due to insufficient number of participants with events. | 6.01 [4.53 to 7.26]
Statistical Analysis 1: Comparison: C1071003 Cohort A vs RWD: Flatiron Health Database; Test type: Other; p = 0.0011, Regression, Cox; Hazard Ratio (HR) = 0.52, 95% CI 2-sided [0.38 to 0.71] — [estimate comment as in outcome 2, analysis 1]

5. Other Pre Specified Outcome: Time to Next Treatment (TTNT): C1071003 Cohort A Versus TM-MM Database Using IPTW Analysis
Description: TTNT: A) C1071003 Cohort A: time from date of first dose of elranatamab to initiation of the next treatment line. Participants were censored at death, loss to or end of follow-up. B) TM-MM Database: time from SOC to start of the next treatment line. Participants were censored at loss to follow-up, death, or end of the study period. Kaplan Meier method was used for analysis. Retrospective data was evaluated in this observational study for approximately 9 months.
Time Frame: C1071003: Date of first dose to start of next treatment line or censoring whichever occurred first (max follow-up of 2.09Y); TM-MM Database: SOC to start of next treatment line or censoring whichever occurred first (max follow-up of 4.22Y)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | C1071003 Cohort A | RWD: TM-MM Database
Number analyzed (Participants) | 118 | 277
Months | NA [4.01 to NA] — Median and upper limit of 95% CI could not be estimated due to insufficient number of participants with events. | 12.06 [11.47 to 14.95]
Statistical Analysis 1: Comparison: C1071003 Cohort A vs RWD: TM-MM Database; Test type: Other; p = 0.503, Regression, Cox; Hazard Ratio (HR) = 0.759, 95% CI 2-sided [0.337 to 1.710] — [estimate comment as in outcome 2, analysis 1]

6. Other Pre Specified Outcome: TTNT: C1071003 Cohort A Versus Flatiron Health Database Using IPTW Analysis
Description: TTNT: A) C1071003 Cohort A: time from date of first dose of elranatamab to initiation of the next treatment line. Participants were censored at death, loss to or end of follow-up. B) Flatiron Health Database: time from SOC to start of the next treatment line. Participants were censored at loss to follow-up, death, or end of the study period. Kaplan Meier method was used for analysis. Retrospective data was evaluated in this observational study for approximately 9 months.
Time Frame: C1071003: Date of first dose to start of next treatment line or censoring whichever occurred first (max follow-up of 2.09Y); Flatiron Health Database: SOC to start of next treatment line or censoring whichever occurred first (max follow-up of 6.45Y)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | C1071003 Cohort A | RWD: Flatiron Health Database
Number analyzed (Participants) | 118 | 238
Months | NA [14.06 to NA] — Median and upper limit of 95% CI could not be estimated due to insufficient number of participants with events. | 7.39 [6.24 to 9.3]
Statistical Analysis 1: Comparison: C1071003 Cohort A vs RWD: Flatiron Health Database; Test type: Other; p < 0.0001, Regression, Cox; Hazard Ratio (HR) = 0.38, 95% CI 2-sided [0.26 to 0.57] — [estimate comment as in outcome 2, analysis 1]

7. Other Pre Specified Outcome: Time to Treatment Discontinuation (TTD): C1071003 Cohort A Versus TM-MM Database Using IPTW Analysis
Description: TTD: A) C1071003 Cohort A: time from the date of first dose of elranatamab to discontinuation. Participants were censored at death, loss to or end of follow-up. B) TM-MM Database: time from initiation of SOC to discontinuation (end) of the SOC. Participants were censored at loss to follow-up, death, or end of the study period. Kaplan Meier method was used for analysis. Retrospective data was evaluated in this observational study for approximately 9 months.
Time Frame: C1071003: Date of first dose to discontinuation or censoring whichever occurred first (max follow-up of 2.09Y); TM-MM Database: SOC to discontinuation of SOC or censoring whichever occurred first (max follow-up of 4.22Y)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | C1071003 Cohort A | RWD: TM-MM Database
Number analyzed (Participants) | 118 | 277
Months | 2.46 [2.04 to 10.19] | 5.59 [4.99 to 7.79]
Statistical Analysis 1: Comparison: C1071003 Cohort A vs RWD: TM-MM Database; Test type: Other; p = 0.706, Regression, Cox; Hazard Ratio (HR) = 0.918, 95% CI 2-sided [0.587 to 1.436] — [estimate comment as in outcome 2, analysis 1]

8. Other Pre Specified Outcome: TTD: C1071003 Cohort A Versus Flatiron Health Database Using IPTW Analysis
Description: TTD: a) C1071003 Cohort A: time from the date of first dose of elranatamab to discontinuation. Participants were censored at death, loss to or end of follow-up. B) Flatiron Health Database: time from initiation of the SOC to discontinuation (end) of the SOC. Participants were censored at loss to follow-up, death, or end of the study period. Kaplan Meier method was used for analysis. Retrospective data was evaluated in this observational study for approximately 9 months.
Time Frame: C1071003: Date of first dose to discontinuation or censoring whichever occurred first (maximum of 2.09Y); Flatiron Health Database: SOC to discontinuation of SOC or censoring whichever occurred first (maximum of 6.45Y)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | C1071003 Cohort A | RWD: Flatiron Health Database
Number analyzed (Participants) | 118 | 238
Months | 6.87 [2.56 to 10.41] | 5.32 [4.17 to 6.64]
Statistical Analysis 1: Comparison: C1071003 Cohort A vs RWD: Flatiron Health Database; Test type: Other; p = 0.0182, Regression, Cox; Hazard Ratio (HR) = 0.68, 95% CI 2-sided [0.52 to 0.88] — [estimate comment as in outcome 2, analysis 1]

ADVERSE EVENTS:
Time Frame: All-cause mortality: During follow-up duration of approximately 25.08 months for C1071003, 50.64 months for RWD: TM-MM database and 77.4 months for RWD: Flatiron Health database; available retrospective data was evaluated in this observational study for approximately 9 months; for adverse events it was not applicable as adverse event data was not planned to be evaluated
Description: This study is retrospective and observational in nature, it involves data that exist as structured data by the time of study start. The minimum criteria for reporting an adverse event (AE) (i.e., identifiable participant, identifiable reporter, a suspect product, and event) cannot be met. Hence, adverse events were not planned to be evaluated and explains 0 at risk.
Arm/Group | C1071003 Cohort A | RWD: TM-MM Database | RWD: Flatiron Health Database
All-Cause Mortality (participants affected / at risk) | 54/118 | 128/277 | 150/238
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
There were some limitations of the study resulting in poor overlap between study arms suggesting that groups are not well comparable in terms of the observed confounding characteristics used for adjustment. This should be taken into consideration when interpreting results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-05-28): https://cdn.clinicaltrials.gov/large-docs/24/NCT06504524/Prot_SAP_000.pdf